CLINICAL TRIAL: NCT01178502
Title: Warfarin Dosing Algorithm for Personalized Warfarin Pharmacotherapy in Korean Patients
Brief Title: PGx Study to Develop and Validate the Predictive Warfarin Dosing Algorithm for Personalized Warfarin Pharmacotherapy
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Other Study IDs: 09-025
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples were taken from patients for genotyping about 8ml
Oversight: Data Monitoring Committee: No

SUMMARY:
To develop and validate the predictive warfarin dosing algorithm.

DETAILED DESCRIPTION:
This study aims to develop and validate the predictive warfarin dosing algorithm for personalized warfarin pharmacotherapy in Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* the patients taking warfarin

Exclusion Criteria:

* noncompliance

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients taking warfarin
Sampling Method: Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To Develop and Validate the Predictive Warfarin Dosing Algorithm | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University, Busan, South Korea